CLINICAL TRIAL: NCT02028312
Title: A Phase IV, Randomized, Parallel Group, Investigator-Masked Evaluation of the Effect of Loteprednol Etabonate Ophthalmic Gel 0.5% on the Initiation of Dry Eye Treatment With Restasis®
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Per Sponsor
Sponsor: Edward Holland, MD (Other)
Responsible Party: Sponsor-Investigator, Edward Holland, MD, Sponsor-Investigator, Holprovision
Organization: Holprovision (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI.HER-002
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Loteprednol Etabonate; Lubricant Eye Drops; Cyclosporins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol etabonate + Restasis (Active Comparator): Loteprednol Etabonate Ophthalmic Gel 0.5%, BID 30 days Restasis, BID 45 days
  Interventions: Drug: Loteprednol etabonate; Drug: Restasis
- Artificial Tears + Restasis (Placebo Comparator): Artificial Tears, BID 30 days Restasis, BID 45 days
  Interventions: Drug: Artificial Tears; Drug: Restasis

INTERVENTIONS:
Drug: Loteprednol etabonate
  Arms: Loteprednol etabonate + Restasis
Drug: Artificial Tears
  Arms: Artificial Tears + Restasis
Drug: Restasis

SUMMARY:
A pilot study to evaluate the impact of Lotemax® Gel (loteprednol etabonate ophthalmic gel 0.5%) on the initiation of Restasis® (cyclosporine ophthalmic emulsion 0.05%) therapy in subjects with dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study-related procedures and provide Health Insurance Portability and Accountability Act (HIPAA) authorization.
2. Are between the ages of 21 and 80 inclusive.
3. Have not worn contact lenses for at least 1 month prior to the study and agrees not to wear contact lenses during the study.
4. Have been on stable oral medications for 1 month prior to the study.
5. Are in generally good and stable overall health.
6. Are a woman of child bearing potential (WOCBP) who is not pregnant or lactating and not sexually active (i.e. abstinent) at Visit 1 and willing to remain so through Visit 4. Alternatively, a WOCBP who is not abstinent must have been using an acceptable method of birth control for at least 4 weeks prior to Visit 1 and throughout the study.
7. Are women who have undergone one of the following sterilization procedures at least 1 month prior to Visit 1:

   1. Bilateral tubal ligation
   2. Hysterectomy
   3. Hysterectomy with unilateral or bilateral oophorectomy.
   4. Bilateral oophorectomy
8. Are likely to comply with the eye drop regime, study guidelines, and study visits.

Exclusion Criteria:

1. Have a history of Stevens-Johnson Syndrome or ocular pemphigoid.
2. Have had punctual plugs inserted or removed; or punctual cautery 3 months prior to Visit 1/Screening and Baseline Visit and throughout the study.
3. Have had intra-ocular surgery within 6 months prior to the Visit 1/Screening and Baseline Visit.
4. Have a history of liver disease.
5. Be pregnant or lactating.
6. Have severe clinical vitamin deficiencies or a history of vitamin overdose.
7. Have a highly variable vitamin intake.
8. Wear contact lenses.
9. Have unstable use of systemic or topical medications known to create dry eye.
10. Have corneal pathology, which could, of itself, cause an ocular surface disorder.
11. Have used glaucoma medications, topical or oral within 30 days of Visit 1/Screening and Baseline Visit.
12. Have unstable diabetes mellitus.
13. Have an allergy or sensitivity to Lotemax® Gel, Restasis®, or non-preservative artificial tears.
14. Have used topical steroids or Restasis® within 1 month prior to the Screening and Baseline Visit and throughout the study, except the study medication provided per the protocol.
15. Have a condition for which steroid use would be contraindicated (e.g. viral infection).
16. Use other topical ocular agents other than tear replacements within 1 week prior to the Screening and Baseline Visit and throughout the study.
17. Have been exposed to an investigational drug within the preceding 30 days.
18. In the opinion of the investigator or study coordinator, be unwilling or unable to comply with the study protocol or unable to successfully instill eye drops.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Fluorescein corneal staining scores | 60 Days

SECONDARY OUTCOMES:
Lissamine green conjunctival staining | 60 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Eye Institute, Edgewood, Kentucky, United States